CLINICAL TRIAL: NCT02809365
Title: The Impact on Quality of Life of Novel Glucose -Sensing Technology Used by Individuals With Type 2 Diabetes on Intensive-insulin Therapy
Brief Title: FreeStyle Libre- Effect on QOL in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, zohar landau, Head of Pediatric Endocrinology Unit, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0096-16-WOMC
Record Dates: First submitted 2016-06-08; First posted 2016-06-22 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes
Keywords: insulin treated
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Libre (Other): FreeStyle Libre users: FreeStyle Libre Flash Glucose Monitoring System is an interstitial glucose monitoring system intended to be replacement for the capillary blood glucose measurement. The system contains several features that distinguish it from exiting sensor technology including no user calibration during 14 days of wear. The sensor is applied to the upper arm of the patient and the hand-held reader is used to scan the sensor to receive glucose result along with historic results with a 15 min frequency for up to 8 hours.
  Interventions: Device: FreeStyle Libre
- SMBG (Other): Self monitoring blood glucose: patients in this arm will measure blood glucose with personal glucometer
  Interventions: Device: personal glucometer

INTERVENTIONS:
Device: FreeStyle Libre — Addition of FreeStyle Libre system for 10 weeks to the treatment of uncontrolled Type 2 diabetic patients currently on multiple daily injections
  Arms: Libre
Device: personal glucometer — Subjects in the Control Group will measure blood glucose levels by personal glucometer (SMBG = self monitoring blood glucose)
  Other Names: SMBG
  Arms: SMBG

SUMMARY:
This is a randomized controlled study in type 2 diabetic patients who are presently uncontrolled on at least 2 injections of insulin daily with an A1C >7.5 % and <10%. Patients need to be stabilized on their MDI for 1 week then randomized to either SBGM or FreeStyle Libre for 10 weeks.

DETAILED DESCRIPTION:
FreeStyle Libre Flash Glucose Monitoring System is an interstitial glucose monitoring system intended to be replacement for the capillary blood glucose measurement. The system contains several features that distinguish it from exiting sensor technology including no user calibration during 14 days of wear. The sensor is applied to the upper arm of the patient and the hand-held reader is used to scan the sensor to receive glucose result along with historic results with a 15 min frequency for up to 8 hours.

An AGP (=Ambulatory Glucose Profile) report is a way to present the glucose data collected by the time of day that has several advantages: demonstrates median glucose levels and the 25-75%, 10-90% excursions as well as the tendency for hypo or hyperglycemia throughout the day. This integration of results gives a more complete picture of the glucose control throughout the week/s while eliminating the "noise" from outliers.

The hypothesis is that the addition of FreeStyle Libre system for 10 weeks to the treatment of uncontrolled Type 2 diabetic patients currently on MDI, will produce a modification of behavior/life style and improvement in treatment satisfaction, quality of life and glycemic control and reduce the number of any/major hypoglycemia events.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes - more than 1 year
2. Age: 30 - 80 yrs
3. Treated with MDI: ≥ 2 injections daily
4. HbA1c: 7.5% to 10%
5. Willing to measure 7 daily blood tests at least one day each week
6. Willing to sign informed consent

Exclusion Criteria:

1. Type 1 diabetes
2. CV event within the last 6 months
3. Steroid therapy > 7 days in last 6 months
4. Retinopathy - grade 3
5. Creatinine >2 mg%

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Improvement of diabetes treatment satisfaction measured by the 'Diabetes Treatment Satisfaction Questionnaire' (DTSQ) | 10 weeks

SECONDARY OUTCOMES:
Improvement of quality of life. | 10 weeks
  This outcome will be measured by a validated diabetes - specific quality of life questionnaire (DQOL).
Assessment of satisfaction from the FreeStyle Libre system | 10 weeks
  This outcome will be measure by a questionnaire developed by the investigators using specific items evaluating the use of the Libre System.
Improvement of HbA1c | 10 weeks
  This outcome will be measured in capillary blood sample.
Percent to reach target HbA1c as defined personally by the physician | 10 weeks
  This outcome will be assessed using the result of the HbA1c.
Reduction in hypoglycemic events <54 mg% | 10 weeks
  By comparing events of glucose levels below 54 mg% in the intervention group versus the control group.
Reduction in hypoglycemic events <70 mg% | 10 weeks
  By comparing events of glucose levels below 70 mg% in the intervention group versus the control group.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - E. Wolfson Medical Center, Holon
  - Wolfson Medical Center, Bariatric Surgery Clinic, Holon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaron M, Roitman E, Aharon-Hananel G, Landau Z, Ganz T, Yanuv I, Rozenberg A, Karp M, Ish-Shalom M, Singer J, Wainstein J, Raz I. Effect of Flash Glucose Monitoring Technology on Glycemic Control and Treatment Satisfaction in Patients With Type 2 Diabetes. Diabetes Care. 2019 Jul;42(7):1178-1184. doi: 10.2337/dc18-0166. Epub 2019 Apr 29. PMID 31036546